# Auditory Brain Training to Enhance Satisfaction and Usage of New Hearing Aids by Older Adults

NCT04230876

Version Date/Number: 6/14/22

## **TABLE OF CONTENTS**

| Α | INT | RODUCTION | 3 |
|---|---|---|---|
| | A1<br>A2 | STUDY ABSTRACT PRIMARY HYPOTHESIS | |
| | A3 | PURPOSE OF THE STUDY PROTOCOL | 4 |
| В | BAC | KGROUND | 4 |
| | B1<br>B2 | PRIOR LITERATURE AND STUDIES RATIONALE FOR THIS STUDY | |
| С | STU | DY OBJECTIVES | 7 |
| | C1 | PRIMARY AIM | 7 |
| | C2 | SECONDARY AIM | |
| _ | C3 | RATIONALE FOR THE SELECTION OF OUTCOME MEASURES | |
| D | | ESTIGATIONAL AGENT | |
| | D1<br>D2 | PRECLINICAL DATA | |
| | D3 | Dose Rationale and Risk/Benefits | |
| Ε | STU | DY DESIGN | 7 |
| | E1 | OVERVIEW OR DESIGN SUMMARY | 7 |
| | E2 | SUBJECT SELECTION AND WITHDRAWAL | 8 |
| | 2.a | Inclusion Criteria | |
| | 2.a<br>2.b | Exclusion Criteria Ethical Considerations | _ |
| | 2.c | Subject Recruitment Plans and Consent Process | |
| | 2.d | Randomization Method and Blinding | |
| | 2.e | Risks and Benefits | 9 |
| | 2.f | Early Withdrawal of Subjects | |
| | 2.g<br>2.h | When and How to Withdraw Subjects | |
| | 2. <i>n</i><br>E3 | Data Collection and Follow-up for Withdrawn Subjects | |
| | 3.a | Description | |
| | 3.b | Treatment Regimen | |
| | 3.c | Method for Assigning Subjects to Treatment Groups | 10 |
| | 3.d | Preparation and Administration of Study Drug | |
| | 3.e | Subject Compliance Monitoring | |
| | 3.f<br>3.g | Prior and Concomitant TherapyPackaging | |
| | 3.y<br>3.h | Blinding of Study Drug | |
| | 3.i | Receiving, Storage, Dispensing and Return | |
| F | STU | DY PROCEDURES | 10 |
| | F1 | Screening for Eligibility | 10 |
| | F2 | SCHEDULE OF MEASUREMENTS | |
| | F3 | VISIT 1 | |
| | F4 | VISIT 2 ETC | |
| | F5<br><i>5.a</i> | Safety and Compliance Monitoring | |
| | 5.b | Medical Monitoring | |
| | i | Investigator only | 11 |
| | ii | Independent expert to monitor | .11 |

| iii Institutional Data and Safety Monitoring Board 11 iv Independent Data and Safety Monitoring Board 11 iv Independent Data and Safety Monitoring Board 11 5 c Definitions of Adverse Events 11 i Relationship 11 ii Severity 11 iii Severity 11 iii Expectedness 11 5 e Data Collection Procedures for Adverse Events 11 5 f Reporting Procedures 12 5 f Report Forus Machana 12 G STATISTICAL PLAN 12 G1 SAMPLE SIZE DETERMINATION AND POWER 12 G2 Interim Monitoring AND EARLY STOPPING 12 G3 ANALYSIS PLAN 12 G4 STATISTICAL METHODS 12 G5 MISSING OUTCOME DATA 12 G6 | _ | | | |
|---|---|---|---|---|
| 5.c Definitions of Adverse Events. 11 5.d Classification of Events. 11 i Relationship. 11 iii Expectedness. 11 5.e Data Collection Procedures for Adverse Events 11 5.f Reporting Procedures. 12 5.g Adverse Event Reporting Period 12 5.h Post-study Adverse Event 12 F6 STUDY OUTCOME MEASUREMENTS AND ASCERTAINMENT 12 G STATISTICAL PLAN. 12 G1 SAMPLE SIZE DETERMINATION AND POWER 12 G2 INTERIM MONITORING AND EARLY STOPPING. 12 G3 ANALYSIS PLAN. 12 G4 STATISTICAL METHODS 12 G5 MISSING OUTCOME DATA. 12 G6 UNBLINDING PROCEDURES. 12 H DATA HANDLING AND RECORD KEEPING 12 H1 CONFIDENTIALITY AND SECURITY 13 H2 TRAINING. 13 H3 CASE REPORT FORMS AND SOURCE DOCUMENTS. 13 H4 RECORDS RETENTION. 13 <t< td=""><td></td><td></td><td></td><td></td></t<> | | | | |
| 5.d Classification of Events. 11 i Relationship 11 ii Seventy 11 iii Expectedness 11 5.e Data Collection Procedures 12 5.f Reporting Procedures 12 5.g Adverse Event Reporting Period 12 5.h Post-study Adverse Event 12 F6 STUDY OUTCOME MEASUREMENTS AND ASCERTAINMENT 12 G STATISTICAL PLAN 12 G1 SAMPLE SIZE DETERMINATION AND POWER 12 G2 INTERIM MONITORING AND EARLY STOPPING 12 G2 INTERIM MONITORING AND EARLY STOPPING 12 G3 ANALYSIS PLAN 12 G4 STATISTICAL METHODS 12 G5 MISSING OUTCOME DATA 12 G6 UNBLINDING PROCEDURES 12 H DATA HANDLING AND RECORD KEEPING 12 H1 CONFIDENTIALITY AND SECURITY 13 H2 TRAINING 13 H3 13 CASE REPORT FORMS AND SOURCE DOCUMENTS 13 <td< th=""><th></th><th></th><th></th><th></th></td<> | | | | |
| Relationship | | | | |
| iii | | 5.u<br>i | | |
| III Expectedness. | | i<br>ii | | |
| 5.e Data Collection Procedures for Adverse Events 11 5.f Reporting Procedures 12 5.g Adverse Event Reporting Period 12 5.h Post-study Adverse Event 12 F6 STUDY OUTCOME MEASUREMENTS AND ASCERTAINMENT 12 G STATISTICAL PLAN 12 G1 SAMPLE SIZE DETERMINATION AND POWER 12 G2 INTERIM MONITORING AND EARLY STOPPING 12 G3 ANALYSIS PLAN 12 G4 STATISTICAL METHODS 12 G5 MISSING OUTCOME DATA 12 G6 UNBLINDING PROCEDURES 12 H DATA HANDLING AND RECORD KEEPING 12 H1 CONFIDENTIALITY AND SECURITY 13 H2 TRAINING 13 H3 CASE REPORT FORMS AND SOURCE DOCUMENTS 13 H4 RECORDS RETENTION 13 H5 PERFORMANCE MONITORING 13 H6 PERFORMANCE MONITORING 13 H1 STUDY MONITORING PLAN 13 H1 STUDY ADMINISTRATION 13 | | | | |
| 5.f Reporting Procedures 12 5.g Adverse Event Reporting Period 12 5.h Post-study Adverse Event 12 F6 STUDY OUTCOME MEASUREMENTS AND ASCERTAINMENT 12 G STATISTICAL PLAN 12 G1 SAMPLE SIZE DETERMINATION AND POWER 12 G2 INTERIM MONITORING AND EARLY STOPPING 12 G3 ANALYSIS PLAN 12 G4 STATISTICAL METHODS 12 G5 MISSING OUTCOME DATA 12 G6 MISSING OUTCOME DATA 12 G6 UNBLINDING PROCEDURES 12 H DATA HANDLING AND RECORD KEEPING 12 H1 CONFIDENTIALITY AND SECURITY 13 H2 TRAINING 13 H3 CASE REPORT FORMS AND SOURCE DOCUMENTS 13 H4 RECORDS RETENTION 13 H5 PERFORMANCE MONITORING 13 H6 STUDY MONITORING, AUDITING, AND INSPECTING 13 I1 STUDY MONITORING PLAN 13 I2 FUNDING SOURCE AND CONFLICTS OF INTEREST 13 < | | | | |
| 5.g Adverse Event Reporting Period 12 5.h Post-study Adverse Event 12 F6 STUDY OUTCOME MEASUREMENTS AND ASCERTAINMENT 12 G STATISTICAL PLAN. 12 G1 SAMPLE SIZE DETERMINATION AND POWER 12 G2 INTERIM MONITORING AND EARLY STOPPING. 12 G2 INTERIM MONITORING AND EARLY STOPPING. 12 G4 STATISTICAL METHODS 12 G5 MISSING OUTCOME DATA. 12 G6 UNBLINDING PROCEDURES. 12 H DATA HANDLING AND RECORD KEEPING. 12 H1 CONFIDENTIALITY AND SECURITY. 13 H2 TRAINING. 13 H3 CASE REPORT FORMS AND SOURCE DOCUMENTS. 13 H4 RECORDS RETENTION. 13 H5 PERFORMANCE MONITORING. 13 I1 STUDY MONITORING, AUDITING, AND INSPECTING. 13 I1 STUDY MONITORING PLAN. 13 I2 FUNDING SOURCE AND CONFLICTS OF INTEREST. 13 J3 COMMITTEES 13 J4 SUBJECT STIPENDS OR PA | | 5.f | | |
| 5.h Post-study Adverse Event 12 F6 STUDY OUTCOME MEASUREMENTS AND ASCERTAINMENT 12 G STATISTICAL PLAN | | 5.q | | |
| F6 STUDY OUTCOME MEASUREMENTS AND ASCERTAINMENT. 12 G STATISTICAL PLAN | | | | |
| G1 SAMPLE SIZE DETERMINATION AND POWER 12 G2 INTERIM MONITORING AND EARLY STOPPING 12 G3 ANALYSIS PLAN 12 G4 STATISTICAL METHODS 12 G5 MISSING OUTCOME DATA 12 G6 UNBLINDING PROCEDURES 12 H DATA HANDLING AND RECORD KEEPING 12 H1 CONFIDENTIALITY AND SECURITY 13 H2 TRAINING 13 H3 CASE REPORT FORMS AND SOURCE DOCUMENTS 13 H4 RECORDS RETENTION 13 H5 PERFORMANCE MONITORING 13 I1 STUDY MONITORING, AUDITING, AND INSPECTING 13 I1 STUDY MONITORING PLAN 13 I2 AUDITING AND INSPECTING 13 J STUDY ADMINISTRATION 13 J3 STUDY ADMINISTRATION 13 J4 SUBJECT STIPENDS OR PAYMENTS 13 J3 COMMITTEES 13 J4 SUBJECT STIPENDS OR PAYMENTS 13 J5 STUDY TIMETABLE 14 K PUBLICATION | | F6 | STUDY OUTCOME MEASUREMENTS AND ASCERTAINMENT | 12 |
| G2 INTERIM MONITORING AND EARLY STOPPING. 12 G3 ANALYSIS PLAN. 12 G4 STATISTICAL METHODS. 12 G5 MISSING OUTCOME DATA. 12 G6 UNBLINDING PROCEDURES. 12 H DATA HANDLING AND RECORD KEEPING. 12 H1 CONFIDENTIALITY AND SECURITY. 13 H2 TRAINING. 13 H3 CASE REPORT FORMS AND SOURCE DOCUMENTS. 13 H4 RECORDS RETENTION. 13 H5 PERFORMANCE MONITORING. 13 I1 STUDY MONITORING, AUDITING, AND INSPECTING. 13 I1 STUDY MONITORING PLAN. 13 I2 AUDITING AND INSPECTING. 13 J STUDY ADMINISTRATION. 13 J1 ORGANIZATION AND PARTICIPATING CENTERS. 13 J2 FUNDING SOURCE AND CONFLICTS OF INTEREST. 13 J3 COMMITTEES. 13 J4 SUBJECT STIPENDS OR PAYMENTS. 13 J5 STUDY TIMETABLE. 14 K PUBLICATION PLAN. 14 <t< th=""><th>G</th><th>STA</th><th>TISTICAL PLAN</th><th>12</th></t<> | G | STA | TISTICAL PLAN | 12 |
| G2 INTERIM MONITORING AND EARLY STOPPING. 12 G3 ANALYSIS PLAN. 12 G4 STATISTICAL METHODS. 12 G5 MISSING OUTCOME DATA. 12 G6 UNBLINDING PROCEDURES. 12 H DATA HANDLING AND RECORD KEEPING. 12 H1 CONFIDENTIALITY AND SECURITY. 13 H2 TRAINING. 13 H3 CASE REPORT FORMS AND SOURCE DOCUMENTS. 13 H4 RECORDS RETENTION. 13 H5 PERFORMANCE MONITORING. 13 I1 STUDY MONITORING, AUDITING, AND INSPECTING. 13 I1 STUDY MONITORING PLAN. 13 I2 AUDITING AND INSPECTING. 13 J STUDY ADMINISTRATION. 13 J1 ORGANIZATION AND PARTICIPATING CENTERS. 13 J2 FUNDING SOURCE AND CONFLICTS OF INTEREST. 13 J3 COMMITTEES. 13 J4 SUBJECT STIPENDS OR PAYMENTS. 13 J5 STUDY TIMETABLE. 14 K PUBLICATION PLAN. 14 <t< th=""><th></th><th>C1</th><th>CAMPLE CIZE DETERMINATION AND DOWER</th><th>12</th></t<> | | C1 | CAMPLE CIZE DETERMINATION AND DOWER | 12 |
| G3 ANALYSIS PLAN 12 G4 STATISTICAL METHODS 12 G5 MISSING OUTCOME DATA 12 G6 UNBLINDING PROCEDURES 12 H DATA HANDLING AND RECORD KEEPING 12 H1 CONFIDENTIALITY AND SECURITY 13 H2 TRAINING 13 H3 CASE REPORT FORMS AND SOURCE DOCUMENTS 13 H4 RECORDS RETENTION 13 H5 PERFORMANCE MONITORING 13 I1 STUDY MONITORING, AUDITING, AND INSPECTING 13 I1 STUDY MONITORING PLAN 13 I2 AUDITING AND INSPECTING 13 J STUDY ADMINISTRATION 13 J1 ORGANIZATION AND PARTICIPATING CENTERS 13 J2 FUNDING SOURCE AND CONFLICTS OF INTEREST 13 J3 COMMITTEES 13 J4 SUBJECT STIPENDS OR PAYMENTS 13 J5 STUDY TIMETABLE 14 K PUBLICATION PLAN 14 L1 TABLES 14 L2 Informed Consent DOCUMENTS | | _ | | |
| G4 STATISTICAL METHODS 12 G5 MISSING OUTCOME DATA 12 G6 UNBLINDING PROCEDURES 12 H DATA HANDLING AND RECORD KEEPING 12 H1 CONFIDENTIALITY AND SECURITY 13 H2 TRAINING 13 H3 CASE REPORT FORMS AND SOURCE DOCUMENTS 13 H4 RECORDS RETENTION 13 H5 PERFORMANCE MONITORING 13 I1 STUDY MONITORING, AUDITING, AND INSPECTING 13 I1 STUDY MONITORING PLAN 13 I2 AUDITING AND INSPECTING 13 J STUDY ADMINISTRATION 13 J STUDY ADMINISTRATION 13 J2 FUNDING SOURCE AND CONFLICTS OF INTEREST 13 J3 COMMITTEES 13 J4 SUBJECT STIPENDS OR PAYMENTS 13 J5 STUDY TIMETABLE 14 K PUBLICATION PLAN 14 L ATTACHMENTS 14 L1 TABLES 14 L2 INFORMED CONSENT DOCUMENTS 14 | | | | |
| G5 MISSING OUTCOME DATA | | | | |
| G6 UNBLINDING PROCEDURES 12 H DATA HANDLING AND RECORD KEEPING 12 H1 CONFIDENTIALITY AND SECURITY 13 H2 TRAINING 13 H3 CASE REPORT FORMS AND SOURCE DOCUMENTS 13 H4 RECORDS RETENTION 13 H5 PERFORMANCE MONITORING 13 I STUDY MONITORING, AUDITING, AND INSPECTING 13 I1 STUDY MONITORING PLAN 13 I2 AUDITING AND INSPECTING 13 J STUDY ADMINISTRATION 13 J STUDY ADMINISTRATION 13 J2 FUNDING SOURCE AND CONFLICTS OF INTEREST 13 J3 COMMITTEES 13 J4 SUBJECT STIPENDS OR PAYMENTS 13 J5 STUDY TIMETABLE 14 K PUBLICATION PLAN 14 L ATTACHMENTS 14 L1 TABLES 14 L2 INFORMED CONSENT DOCUMENTS 14 L3 PATIENT EDUCATION BROCHURES 14 L4 SPECIAL PROCEDURES PROTOCOLS < | | | | |
| H DATA HANDLING AND RECORD KEEPING 12 H1 CONFIDENTIALITY AND SECURITY 13 H2 TRAINING | | | | |
| H1 CONFIDENTIALITY AND SECURITY 13 H2 TRAINING 13 H3 CASE REPORT FORMS AND SOURCE DOCUMENTS 13 H4 RECORDS RETENTION 13 H5 PERFORMANCE MONITORING 13 I STUDY MONITORING, AUDITING, AND INSPECTING 13 I1 STUDY MONITORING PLAN 13 I2 AUDITING AND INSPECTING 13 J STUDY ADMINISTRATION 13 J1 ORGANIZATION AND PARTICIPATING CENTERS 13 J2 FUNDING SOURCE AND CONFLICTS OF INTEREST 13 J3 COMMITTEES 13 J4 SUBJECT STIPENDS OR PAYMENTS 13 J5 STUDY TIMETABLE 14 K PUBLICATION PLAN 14 L1 TABLES 14 L2 INFORMED CONSENT DOCUMENTS 14 L3 PATIENT EDUCATION BROCHURES 14 L4 SPECIAL PROCEDURES PROTOCOLS 14 L5 QUESTIONNAIRES OR SURVEYS 14 | | | | |
| H2 TRAINING 13 H3 CASE REPORT FORMS AND SOURCE DOCUMENTS 13 H4 RECORDS RETENTION 13 H5 PERFORMANCE MONITORING 13 I STUDY MONITORING, AUDITING, AND INSPECTING 13 I1 STUDY MONITORING PLAN 13 I2 AUDITING AND INSPECTING 13 J STUDY ADMINISTRATION 13 J1 ORGANIZATION AND PARTICIPATING CENTERS 13 J2 FUNDING SOURCE AND CONFLICTS OF INTEREST 13 J3 COMMITTEES 13 J4 SUBJECT STIPENDS OR PAYMENTS 13 J5 STUDY TIMETABLE 14 K PUBLICATION PLAN 14 L ATTACHMENTS 14 L1 TABLES 14 L2 Informed consent documents 14 L3 Patient education brochures 14 L4 Special procedures protocols 14 L5 Questionnaires or surveys 14 | Н | DAT | | |
| H3 CASE REPORT FORMS AND SOURCE DOCUMENTS 13 H4 RECORDS RETENTION 13 H5 PERFORMANCE MONITORING 13 I STUDY MONITORING, AUDITING, AND INSPECTING 13 I1 STUDY MONITORING PLAN 13 I2 AUDITING AND INSPECTING 13 J STUDY ADMINISTRATION 13 J1 ORGANIZATION AND PARTICIPATING CENTERS 13 J2 FUNDING SOURCE AND CONFLICTS OF INTEREST 13 J3 COMMITTEES 13 J4 SUBJECT STIPENDS OR PAYMENTS 13 J5 STUDY TIMETABLE 14 K PUBLICATION PLAN 14 L ATTACHMENTS 14 L1 TABLES 14 L2 INFORMED CONSENT DOCUMENTS 14 L3 PATIENT EDUCATION BROCHURES 14 L4 SPECIAL PROCEDURES PROTOCOLS 14 L5 QUESTIONNAIRES OR SURVEYS 14 | | H1 | | |
| H4 RECORDS RETENTION 13 H5 PERFORMANCE MONITORING 13 I STUDY MONITORING, AUDITING, AND INSPECTING 13 I1 STUDY MONITORING PLAN 13 I2 AUDITING AND INSPECTING 13 J STUDY ADMINISTRATION 13 J1 ORGANIZATION AND PARTICIPATING CENTERS 13 J2 FUNDING SOURCE AND CONFLICTS OF INTEREST 13 J3 COMMITTEES 13 J4 SUBJECT STIPENDS OR PAYMENTS 13 J5 STUDY TIMETABLE 14 K PUBLICATION PLAN 14 L ATTACHMENTS 14 L1 TABLES 14 L2 Informed Consent documents 14 L3 PATIENT EDUCATION BROCHURES 14 L4 Special procedures protocols 14 L5 QUESTIONNAIRES OR SURVEYS 14 | | | | |
| H5 PERFORMANCE MONITORING 13 I STUDY MONITORING, AUDITING, AND INSPECTING 13 I1 STUDY MONITORING PLAN 13 I2 AUDITING AND INSPECTING 13 J STUDY ADMINISTRATION 13 J1 ORGANIZATION AND PARTICIPATING CENTERS 13 J2 FUNDING SOURCE AND CONFLICTS OF INTEREST 13 J3 COMMITTEES 13 J4 SUBJECT STIPENDS OR PAYMENTS 13 J5 STUDY TIMETABLE 14 K PUBLICATION PLAN 14 L ATTACHMENTS 14 L1 TABLES 14 L2 Informed Consent Documents 14 L3 PATIENT EDUCATION BROCHURES 14 L4 Special procedures protocols 14 L5 Questionnaires or surveys 14 | | | | |
| I STUDY MONITORING, AUDITING, AND INSPECTING 13 11 STUDY MONITORING PLAN. 13 12 AUDITING AND INSPECTING 13 J STUDY ADMINISTRATION 13 J1 ORGANIZATION AND PARTICIPATING CENTERS 13 J2 FUNDING SOURCE AND CONFLICTS OF INTEREST 13 J3 COMMITTEES 13 J4 SUBJECT STIPENDS OR PAYMENTS 13 J5 STUDY TIMETABLE 14 K PUBLICATION PLAN 14 L ATTACHMENTS 14 L1 TABLES 14 L2 INFORMED CONSENT DOCUMENTS 14 L3 PATIENT EDUCATION BROCHURES 14 L4 SPECIAL PROCEDURES PROTOCOLS 14 L5 QUESTIONNAIRES OR SURVEYS 14 | | | | |
| 11 STUDY MONITORING PLAN | | H5 | PERFORMANCE MONITORING | 13 |
| 12 AUDITING AND INSPECTING | I | | | |
| J STUDY ADMINISTRATION 13 J1 ORGANIZATION AND PARTICIPATING CENTERS 13 J2 FUNDING SOURCE AND CONFLICTS OF INTEREST 13 J3 COMMITTEES 13 J4 SUBJECT STIPENDS OR PAYMENTS 13 J5 STUDY TIMETABLE 14 K PUBLICATION PLAN 14 L ATTACHMENTS 14 L1 TABLES 14 L2 INFORMED CONSENT DOCUMENTS 14 L3 PATIENT EDUCATION BROCHURES 14 L4 SPECIAL PROCEDURES PROTOCOLS 14 L5 QUESTIONNAIRES OR SURVEYS 14 | | 11 S | FUDY MONITORING PLAN | 13 |
| J1 ORGANIZATION AND PARTICIPATING CENTERS 13 J2 FUNDING SOURCE AND CONFLICTS OF INTEREST 13 J3 COMMITTEES 13 J4 SUBJECT STIPENDS OR PAYMENTS 13 J5 STUDY TIMETABLE 14 K PUBLICATION PLAN 14 L ATTACHMENTS 14 L1 TABLES 14 L2 INFORMED CONSENT DOCUMENTS 14 L3 PATIENT EDUCATION BROCHURES 14 L4 SPECIAL PROCEDURES PROTOCOLS 14 L5 QUESTIONNAIRES OR SURVEYS 14 | | I2 Au | JDITING AND INSPECTING | 13 |
| J1 ORGANIZATION AND PARTICIPATING CENTERS 13 J2 FUNDING SOURCE AND CONFLICTS OF INTEREST 13 J3 COMMITTEES 13 J4 SUBJECT STIPENDS OR PAYMENTS 13 J5 STUDY TIMETABLE 14 K PUBLICATION PLAN 14 L ATTACHMENTS 14 L1 TABLES 14 L2 INFORMED CONSENT DOCUMENTS 14 L3 PATIENT EDUCATION BROCHURES 14 L4 SPECIAL PROCEDURES PROTOCOLS 14 L5 QUESTIONNAIRES OR SURVEYS 14 | | etii | DV ADMINISTRATION | 12 |
| J2 FUNDING SOURCE AND CONFLICTS OF INTEREST 13 J3 COMMITTEES 13 J4 SUBJECT STIPENDS OR PAYMENTS 13 J5 STUDY TIMETABLE 14 K PUBLICATION PLAN 14 L ATTACHMENTS 14 L1 TABLES 14 L2 INFORMED CONSENT DOCUMENTS 14 L3 PATIENT EDUCATION BROCHURES 14 L4 SPECIAL PROCEDURES PROTOCOLS 14 L5 QUESTIONNAIRES OR SURVEYS 14 | J | | | |
| J3 COMMITTEES 13 J4 SUBJECT STIPENDS OR PAYMENTS 13 J5 STUDY TIMETABLE 14 K PUBLICATION PLAN 14 L ATTACHMENTS 14 L1 TABLES 14 L2 Informed consent documents 14 L3 Patient education brochures 14 L4 Special procedures protocols 14 L5 Questionnaires or surveys 14 | | | | |
| J4 SUBJECT STIPENDS OR PAYMENTS 13 J5 STUDY TIMETABLE 14 K PUBLICATION PLAN 14 L ATTACHMENTS 14 L1 TABLES 14 L2 Informed Consent documents 14 L3 Patient education brochures 14 L4 Special procedures protocols 14 L5 Questionnaires or surveys 14 | | | | |
| J5 STUDY TIMETABLE 14 K PUBLICATION PLAN 14 L ATTACHMENTS 14 L1 TABLES 14 L2 Informed Consent documents 14 L3 Patient education brochures 14 L4 Special procedures protocols 14 L5 Questionnaires or surveys 14 | | | | |
| K PUBLICATION PLAN 14 L ATTACHMENTS 14 L1 TABLES 14 L2 Informed consent documents 14 L3 PATIENT EDUCATION BROCHURES 14 L4 SPECIAL PROCEDURES PROTOCOLS 14 L5 QUESTIONNAIRES OR SURVEYS 14 | | | | |
| L ATTACHMENTS 14 L1 TABLES 14 L2 Informed consent documents 14 L3 Patient education brochures 14 L4 Special procedures protocols 14 L5 Questionnaires or surveys 14 | | J5 S | rudy Timetable | 14 |
| L1 TABLES 14 L2 INFORMED CONSENT DOCUMENTS 14 L3 PATIENT EDUCATION BROCHURES 14 L4 SPECIAL PROCEDURES PROTOCOLS 14 L5 QUESTIONNAIRES OR SURVEYS 14 | K | PUB | LICATION PLAN | 14 |
| L2INFORMED CONSENT DOCUMENTS14L3PATIENT EDUCATION BROCHURES14L4SPECIAL PROCEDURES PROTOCOLS14L5QUESTIONNAIRES OR SURVEYS14 | L | ATT | ACHMENTS | 14 |
| L2INFORMED CONSENT DOCUMENTS14L3PATIENT EDUCATION BROCHURES14L4SPECIAL PROCEDURES PROTOCOLS14L5QUESTIONNAIRES OR SURVEYS14 | | I 1 | TARI ES | 14 |
| L3 PATIENT EDUCATION BROCHURES | | | | |
| L4 SPECIAL PROCEDURES PROTOCOLS 14 L5 QUESTIONNAIRES OR SURVEYS 14 | | | | |
| L5 QUESTIONNAIRES OR SURVEYS | | | | |
| | M | - | | |

## A Introduction

A1 Study Abstract

Auditory training as the potential to dramatically affect older persons' adjustment to a new hearing aid and to maximize the benefits they receive from wearing one. In turn, by wearing hearing aids, they experience easier and more successful communication patterns. They enhance their ability to engage in everyday conversations and will be able to become more socially involved with their family and friends. In this study we will try to determine the extent to which web-based clEAR auditory brain training, with concomitant support from a clEAR in-house audiologist, affects satisfaction with new hearing aids and increases daily use time. Thirty adults over the age of 60 years will receive new hearing aids for the first time. After an adjustment period, half will complete clEAR's auditory brain training program right away and the other half will complete it after a delay period, and both will complete a control condition. To establish the level of feasibility and clinical utility we will measure hearing aid satisfaction, benefit ratings, and hearing aid use time.

### A2 Primary Hypothesis

Use of the web-based cIEAR auditory brain training system with concomitant support from a cIEAR in-house audiologist improves satisfaction with new hearing aids and increases daily use time.

#### A3 Purpose of the Study Protocol

Determine the extent to which web-based cIEAR auditory brain training with concomitant support from a cIEAR in-house audiologist affects satisfaction with new hearing aids and increases daily use time.

## **B** Background

#### **B1** Prior Literature and Studies

Barcroft, J., Sommers, M., Tye-Murray, N., Mauzé, E., Schroy, C., & Spehar, B. (2011). Tailoring auditory training to patient needs with single and multiple talkers: Transfer-appropriate gains on a four-choice discrimination test. International Journal of Audiology, 50(11), 1802–1808.

Barcroft, J., Spehar, B., Tye-Murray, N., & Sommers, M. (2016). Task-and talker-specific gains in auditory training. Journal of Speech, Language, and Hearing Research, 59(4), 862-870.

Sommers, M. S., Tye-Murray, N., Barcroft, J., & Spehar, B. (2015). The effects of meaning-based auditory training on behavioral measures of perceptual effort in individuals with impaired hearing. Seminars in Hearing, 36(4), 263-272.

Tye-Murray, N., Sommers, M., Mauzé, E., Schroy, C., Barcroft, J., & Spehar, B. (2012). Using patient perceptions of relative benefit ad enjoyment to assess auditory training. Journal of the American Academy of Audiology, 23(8), 623–634.

Tye-Murray, N., Spehar, B., Sommers, M., & Barcroft, J. (2016). Auditory training with frequent communication partners. Journal of Speech, Language, and Hearing Research, 59(4), 871-875.

Tye-Murray, N., Spehar, B., Barcroft, J., & Sommers, M. (2017). Auditory training for adults who have hearing loss: A comparison of spaced versus massed practice schedules. Journal of Speech, Language, and Hearing Research, 60(8), 2337-2345.

#### **B2** Rationale for this Study

clEAR auditory brain training has been shown to be effective and that patients like the contact with an audiologist during training. Barcroft et al. (2011; see also Tye-Murray et al., 2017) showed that computerized, game-like auditory training is beneficial for older adults (mean age=66 years, SD=16) who have hearing loss by conducting a 3-year large-scale study that addressed the effectiveness of computerized training for a talker trained with and for a talker not trained with. We also considered whether benefits were maintained three months later. A one-way ANOVA revealed a significant overall effect of training regardless of the talker. In a second study, Adults with hearing loss completed the clEAR program and were placed in a group that trained on either multiple talkers or a single talker (Barcroft et al., 2016). A control group also completed 12 hours of training in American Sign Language. The experimental group's training included a 4-choice discrimination task but not an open-set sentence test. The assessment phase included the same 4-Improvement on 4-choice discrimination was

observed in the experimental group as compared with the control group. Gains were (a) highest when the task and talker were the same between training and assessment; (b) second highest when the task was the same but the talker only partially so; and (c) third highest when task and talker were different. The findings support applications of transfer-appropriate processing to auditory training and favor tailoring programs toward the specific needs of the individuals being trained for tasks, talkers, and perhaps, for stimuli, in addition to other factors.

Auditory brain training has been shown to reduce perceptual effort. Sommers et al. (2015) assessed the extent to which engaging in gamified auditory training would reduce perceptual or listening effort. As the name implies, perceptual effort pertains to the cognitive resources that must be allocated to recognizing speech. Perceptual effort was assessed using an n-back memory task. Eighty-three participants heard lists of words presented without background noise and were asked to continually update their memory of the three most recently presented words. Perceptual effort was gauged by memory for items in the three-back position immediately before, immediately after, and 3 months after participants completed 12 sessions (approximately 8 hours) of the clEAR auditory brain training games. Immediate post-training measures of perceptual effort indicated that participants could remember approximately one additional word compared to pre-training. Moreover, some training gains were retained at the 3-month followup, as indicated by significantly greater recall for the three-back item at the 3month measurement than at pretest. A significant correlation was found between gains in intelligibility and gains in perceptual effort.

Auditory brain training enhances recognition of familiar voices. Tye-Murray et al. (2016) conducted a study to determine whether auditory training with the speech of an adult's spouse would lead to enhanced recognition of that person's speech. Ten older participants (mean age=73 years, SD=6) completed 6 weeks (12 hours) of training. Their spouses recorded the stimuli and each participant (partner with hearing loss) completed auditory training that presented the recordings. Training led participants to better discriminate their spouse's speech, as indicated by the 4-AFC. Subjectively, responses on a questionnaire indicated that training reduced participants' communication difficulties. Couples had been married an average of 14 years showed that providing training with a formerly unfamiliar talker led to significant gains in participants' ability to recognize the speech of the talker, and that gains were seen for the speech of untrained talkers, although not to the same extent.

Patients want regular contact with an audiologist. In a study of 93 adults (mean age=66 years, SD=17), we asked the question, what did you like best about the auditory training (Tye-Murray et al., 2012). One of the three top answers was "regular contact with an audiologist". The other two were "the games were fun to play" and "training gave me empowerment over my hearing loss." By completing auditory brain training, participants also reported increased confidence to engage in everyday conversations.

## C Study Objectives

#### C1 Primary Aim

It is the objective of this study to determine if the use of clEAR following a first-time hearing aid fitting will increase satisfaction and daily hearing aid use.

#### C2 Secondary Aim

Ν'Α

#### C3 Rationale for the Selection of Outcome Measures

- 1. Primary outcome measures are questionnaires used in hearing clinics to assess hearing aid satisfaction.
- 2. Hearing aids log use time. This information will also be collected to determine the average daily use time for each participant.

## **D** Investigational Agent

D1 Preclinical Data

N/A

D2 Clinical Data to Date

N/A

D3 Dose Rationale and Risk/Benefits

N/A

## E Study Design

## E1 Overview or Design Summary

All qualified participants will first be fitted with one hearing aid using manufacturer recommended settings. The settings will be verified using real-ear measurements and any initial adjustments to the hearing aid will be made at the time of fitting. The participants will return again in 2-3 weeks to complete any final adjustments needed before they continue with the protocol.

After fitting and final adjustments are complete, all participants will be receive aided speech perception testing using the Speech in Noise Test (SPIN) and the NU-6.

Half of the participants will be assigned to the Early Group and receive 8 hours of clEAR auditory brain training in 20 minute intervals spread over four weeks. The other half will be assigned to the Late Group and receive the clEAR training after

a four week control period. The Early Group will do the control period after their training period.

For the control period, participants will be given a choice of three audio books stored on Amazon Kindle (a mystery, a biography, or a popular fiction) to ensure that the book will engage a participant's interest and that they will be motivated to follow the training schedule. They will be provided with a formal schedule that parallels the training schedule for the cIEAR training, and will receive 8 hours of training. We will confirm their compliance through weekly phone calls, email, and by asking them to report how far along they are in the book. If participants do not have a tablet for reading, they will provided with a loaner tablet which allow access to Kindle books. A final period will be four weeks after either type of intervention.

At the end of each period participants will receive the speech perception battery (SPIN and NU-6) and the subjective assessment battery includes questionnaires and scales commonly used to assess hearing aid satisfaction and changes in listening challenges. The battery will include three subjective measures, The SADL (Satisfaction with Amplification in Daily Life), the IOI-HA (The International Outcome Inventory for Hearing Aids, and the COSI (Client Oriented Scale of Improvement). Finally, at the end of the clEAR training period participants will complete a questionnaire designed to gain feedback about the games, participants will also complete a questionnaire about their clEAR experience, indicating what they did and did not like about the system.

#### E2 Subject Selection and Withdrawal

#### 2.a Inclusion Criteria

All participants have the same inclusion/exclusion criteria but be assigned to one of two groups that differ only in the schedule, this will allow participants will act as their own control group.

All participants will:

- 1. Be over 60 years old
- 2. Have a bilateral sensorineural hearing loss mild-to-severe range
- 3. Vision will need to be corrected to at least 20/40 so participants can see the training games on the computer or tablet monitor.

#### 2.a Exclusion Criteria

English must be the first language of the participant
Participants must pass a dementia screener (MMSE)
Must have the manual dexterity to manipulate and insert a hearing aid
Must have an email address and access to the internet

2.b Ethical Considerations

# Nobody will be discriminated against based on conditions not noted in the inclusion/exclusion criteria.

#### 2.c Subject Recruitment Plans and Consent Process

Lists of potential participants will be obtained from multiple sources including the Washington University's Volunteers for Health program and from an extensive database maintained in the Tye-Murray lab. Potential participants will hear about the study and complete a health and hearing screening questionnaire over the telephone. If they pass the telephone screening, they will be asked to come to the hearing lab for the hearing and vision assessment. The hearing screening will include pure-tone threshold testing and speech perception testing at comfortable levels.

To be enrolled in the study potential participants will have bilateral mild to severe sensori-neural hearing loss, and have never used hearing aids. They will also require the basic skills for wearing and maintaining a hearing aid including the manual dexterity to insert the aid and the anatomy required to wear the aid. They will also have corrected static visual acuity of 20/40 or better. They will be required to pass a dementia screener (MMSE). If they qualify for the study and wish to continue they will be consented after completing the assessments. Those that do not qualify will be paid for their time and any collected data destroyed.

#### 2.d Randomization Method and Blinding

Because participants act as their own control per se, they will not be randomized and no blinding will occur.

#### 2.e Risks and Benefits

There are no foreseeable risks to the participant beyond the basic risks associated with hearing aid fitting. These risks are rare but include possible skin irritation from the device or the occasional uncomfortably loud sound. Hearing aids are equipped with safety mechanisms that are supposed to reduce the possibility that a very uncomfortable level is produced.

The participant will participate in a study that provides amplification and auditory training. These devices and procedures are designed to be of benefit to individuals with hearing loss. The participants will also be providing feedback on their experiences. This feedback may improve the procedures and methods currently used in online auditory training practices, this may benefit society.

#### 2.f Early Withdrawal of Subjects

Participants that have not completed the study but can no longer participate will be asked to return the hearing aid. They will be reimbursed for their time at 10\$/hour.

#### 2.g When and How to Withdraw Subjects

If it is deemed that they can no longer fulfill the needs of the study because they are not training or coming to the in-clinic assessments participants will be notified by phone or email if they are to be withdrawn from the study.

#### 2.h Data Collection and Follow-up for Withdrawn Subjects

There will be no follow-up with withdrawn participants.

| E3 | Study | Drug |
|----|-------|------|
|----|-------|------|

3.a Description

N/A

3.b Treatment Regimen

N/A

3.c Method for Assigning Subjects to Treatment Groups

N/A

3.d Preparation and Administration of Study Drug

N/A

3.e Subject Compliance Monitoring

N/A

3.f Prior and Concomitant Therapy

N/A

3.g Packaging

N/A

3.h Blinding of Study Drug

N/A

3.i Receiving, Storage, Dispensing and Return

N/A

#### F Study Procedures

#### F1 Screening for Eligibility

A telephone survey will screen all potential participants that would not be eligible for reasons other than the hearing and vision screening. Hearing and vision testing will be conducted after the informed consent process.

#### F2 Schedule of Measurements

| F3 | Visit 1 |
|-----|------------------------------------------------|
| F4 | Visit 2 etc. |
| F5 | Safety and Adverse Events |
| 5.a | Safety and Compliance Monitoring |
| 5.b | Medical Monitoring |
| i | Investigator only |
| ii | Independent expert to monitor |
| iii | Institutional Data and Safety Monitoring Board |
| iv | Independent Data and Safety Monitoring Board |
| 5.c | Definitions of Adverse Events |
| 5.d | Classification of Events |
| i | Relationship |
| ii | Severity |
| iii | Expectedness |
| 5.e | Data Collection Procedures for Adverse Events |

#### 5.f Reporting Procedures

- 5.g Adverse Event Reporting Period
- 5.h Post-study Adverse Event
- F6 Study Outcome Measurements and Ascertainment

#### **G** Statistical Plan

#### G1 Sample Size Determination and Power

We determined the power to detect an effect size for differences as large as or larger than in Tye-Murray et al. (mean = .733, SD = .783) with an alpha level of .05 will exceed .95 using a one-tailed test for the within-subjects comparisons in each group.

#### G2 Interim Monitoring and Early Stopping

We will monitor progress in the software to be sure participants are following protocol.

#### G3 Analysis Plan

We will assess the effect of training on hearing aid use time, changes in speech perception, and subjective changes indicated by the questionnaire rating-scale responses. Three post-fitting times will be assessed to look at the effects of clEAR testing (Baseline/post-fitting, post-training, post control, and four weeks post intervention).

#### G4 Statistical Methods

Data will be analyzed with t-tests and repeated measures ANOVA.

## G5 Missing Outcome Data

Participants with missing data will not be included in the analyses for that outcome measure.

## **G6** Unblinding Procedures

N/A

## H Data Handling and Record Keeping

| H1 | Confidentiality and Security |
|---|---|
| Н2 | Training |
| НЗ | Case Report Forms and Source Documents |
| Н4 | Records Retention |
| Н5 | Performance Monitoring |
| 1 ; | Study Monitoring, Auditing, and Inspecting |
| <i>I1</i> | Study Monitoring Plan |
| 12 | Auditing and Inspecting |
| | Study Administration |
| | Study Administration |
| J1 | Organization and Participating Centers |
| J2 | Funding Source and Conflicts of Interest |
| | UDE INFO FROM CIRC? BUT WE ARE NOT THE PI, SO IT WOULDN'T MAKE SE HERE. |
| J3 | Committees |
| <b>J4</b><br>Parti | Subject Stipends or Payments icipants will be paid \$10/hour for the time spent in assessments and training. |

Other - The project involves first time hearing aid users. We need to control for the level of technology and hearing aid quality across participants, so the hearing aid will be provided. The aid will be 'used' after the study so the participant will be allowed to keep the aid after the study is complete.

#### J5 Study Timetable

## **K** Publication Plan

### L Attachments

#### L1 Tables

#### L2 Informed consent documents

| Adult SBIR HA and AT Informed | Consent & Assent | 1 | 407 k | Ε | 08/20/19 |
|-------------------------------|------------------|---|-------|---|----------|
| consent.rtf | Forms | | | | |

#### L3 Patient education brochures

## L4 Special procedures protocols

#### L5 Questionnaires or surveys

| Attachment Name | Category | Ver | Size | | Attached |
|---|---|---|---|---|---|
| JIT Letter.doc | Notice of Just in Time (JIT) Documentation | 1 | 25 k | Е | 08/15/19 |
| <u>Telephone</u> | Recruitment Script: Phone | 1 | 59 k | Е | 08/19/19 |

| Questionnaire.rtf | | | | | |
|---|---|---|---|---|---|
| AT and HA Flier.rtf | Recruitment Materials:<br>Ads/Brochures/Posters/News<br>Release/Fliers | 1 | 115 k | Е | 08/19/19 |
| COSI.pdf | Subject Data Collection<br>Instruments | 1 | 36 k | Е | 08/21/19 |
| Demographic - Case History Form.rtf | Subject Data Collection Instruments | 1 | 86 k | Е | 08/20/19 |
| Email and Phone Script for Followups.doc | Subject Data Collection<br>Instruments | 1 | 23 k | Е | 08/20/19 |
| IOI-HA.pdf | Subject Data Collection<br>Instruments | 1 | 37 k | Е | 08/21/19 |
| SADL Form.pdf | Subject Data Collection Instruments | 1 | 58 k | Е | 08/21/19 |
| Assurance Form Signed.pdf | Assurance Document | 1 | 226 k | E | 08/21/19 |

#### **M** References

Barcroft, J., Sommers, M., Tye-Murray, N., Mauzé, E., Schroy, C., & Spehar, B. (2011). Tailoring auditory training to patient needs with single and multiple talkers: Transfer-appropriate gains on a four-choice discrimination test. International Journal of Audiology, 50(11), 1802–1808.

Barcroft, J., Spehar, B., Tye-Murray, N., & Sommers, M. (2016). Task-and talker-specific gains in auditory training. Journal of Speech, Language, and Hearing Research, 59(4), 862-870.

Sommers, M. S., Tye-Murray, N., Barcroft, J., & Spehar, B. (2015). The effects of meaning-based auditory training on behavioral measures of perceptual effort in individuals with impaired hearing. Seminars in Hearing, 36(4), 263-272.

Tye-Murray, N., Sommers, M., Mauzé, E., Schroy, C., Barcroft, J., & Spehar, B.

(2012). Using patient perceptions of relative benefit ad enjoyment to assess auditory training. Journal of the American Academy of Audiology, 23(8), 623–634.

Tye-Murray, N., Spehar, B., Sommers, M., & Barcroft, J. (2016). Auditory training with frequent communication partners. Journal of Speech, Language, and Hearing Research, 59(4), 871-875.

Tye-Murray, N., Spehar, B., Barcroft, J., & Sommers, M. (2017). Auditory training for adults who have hearing loss: A comparison of spaced versus massed practice schedules. Journal of Speech, Language, and Hearing Research, 60(8), 2337-2345.